CLINICAL TRIAL: NCT00441142
Title: Phase I/II Study of ZD6474 (Vandetanib) With Radiation Therapy and Concomitant and Adjuvant Temozolomide in Patients With Newly-Diagnosed Glioblastoma
Brief Title: Zactima With Temodar During Radiation Treatment for Newly Diagnosed Stage IV Brain Tumors
Acronym: Zactima
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Patrick Y. Wen, MD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); University of Virginia (Other); Memorial Sloan Kettering Cancer Center (Other); Henry Ford Hospital (Other)
Responsible Party: Sponsor-Investigator, Patrick Y. Wen, MD, Director, Center For Neuro-Oncology, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-377; IRUSZACT0018 (Other: AstraZeneca)
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma Multiforme; Gliosarcoma
Keywords: Newly diagnosed malignant brain tumors.
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — vandetanib; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase II: Arm A (Control Group: RT + TMZ) (Active Comparator): The "Induction" Phase:
  Temozolomide (75 mg/m2 daily for 6 weeks) with concurrent fractionated radiation therapy for approximately 6 weeks (XRT must be given by external beam to a partial brain field in daily fractions of 180-200 cGy, to a planned total dose to the tumor of approximately 6000 cGy), followed by 4-6 weeks rest.
  Followed by the "Maintenance" Phase:
  12 cycles of adjuvant temozolomide [at 150 mg/m2/day orally for 5 days (days 1-5) of a 28-day TMZ cycle; if 150 mg/m2/day is tolerated without difficulty and the investigator feels the patient can tolerate 200 mg/m2/day, then an increase to a maximum of 200 mg/m2/day for five days every 28 days may be given].
  Interventions: Drug: temozolomide; Radiation: Radiation Therapy
- Phase I + Phase II: Arm B (RT + TMZ + Vandetanib) (Experimental): The "Induction" Phase:
  ZD6474 (Vandetanib) daily (to begin 5-7 days prior to starting participant's RT) Temozolomide (75 mg/m2 daily for 6 weeks) with concurrent fractionated radiation therapy for approximately 6 weeks (XRT must be given by external beam to a partial brain field in daily fractions of 180-200 cGy, to a planned total dose to the tumor of approximately 6000 cGy), followed by 4-6 weeks rest.
  Followed by the "Maintenance" Phase:
  12 cycles of adjuvant temozolomide [at 150 mg/m2/day orally for 5 days (days 1-5) of a 28-day TMZ cycle; if 150 mg/m2/day is tolerated without difficulty and the investigator feels the patient can tolerate 200 mg/m2/day, then an increase to a maximum of 200 mg/m2/day for five days every 28 days may be given].
  ZD6474 (Vandetanib) daily for the twelve (12) 28-day cycles of adjuvant temozolomide, with the option to continue until participant experiences an unacceptable toxicity or his/her tumor progresses.
  Interventions: Drug: ZD6474; Drug: temozolomide; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: ZD6474 — Taken orally once a day (at 100 mg/day is the phase II dose; the MTD determined by the phase I portion of the trial) until disease gets worse or participants experience unacceptable side effects
  Other Names: Vandetanib; Zactima
  Arms: Phase I + Phase II: Arm B (RT + TMZ + Vandetanib)
Drug: temozolomide — During the 'Induction' phase: 75/mg/m2/day temozolomide will be given orally daily for 6 weeks (42 days) during radiation therapy, beginning either the night before or on the first day of the first fraction of radiation, including weekends and holidays. This is followed by a 4-6 week break.
  During the 'Maintenance' phase: The first post-radiation temozolomide cycle will be administered at 150 mg/m2/day orally for 5 days (days 1-5) of a 28-day TMZ cycle. If 150 mg/m2/day is tolerated without difficulty and the investigator feels the patient can tolerate 200 mg/m2/day, then an increase to a maximum of 200 mg/m2/day for five days every 28 days may be given. This is given for 12 cycles.
  Other Names: Temodar
Radiation: Radiation Therapy — Radiotherapy must be given by external beam to a partial brain field in daily fractions of 180-200 cGy, to a planned total dose to the tumor of approximately 6000 cGy.
  Other Names: RT; XRT

SUMMARY:
Phase I:

The purpose of this research study is to determine the safety of the combination treatment of ZD6474 (Vandetanib) with the standard therapy for glioblastomas and gliosarcomas, temozolomide (Temodar) and radiation therapy. This agent is investigational for the treatment of glioblastomas. We will determine the highest dose of ZD6474 (Vandetanib) that can be given safely when combined with temozolomide (Temodar) and radiation therapy.

Phase II:

The purpose of this research study is to determine the efficacy of the combination treatment of ZD6474 (Vandetanib) with the standard therapy for glioblastomas and gliosarcomas, temozolomide (Temodar) and radiation therapy. This agent is investigational for the treatment of glioblastomas.

All subjects participating in this research study must NOT be taking a certain type of anti-seizure medication called enzyme inducing anticonvulsant drugs. These drugs include (but are not limited to) the following medications: Dilantin, Tegretol, Phenobarbital and trileptal.

DETAILED DESCRIPTION:
Currently the standard treatment for glioblastomas and gliosarcomas is temozolomide (Temodar) and radiation therapy. This study is being done because research has shown that glioblastomas have genetic changes that may cause an excess of certain cell growth factors and their receptors, which can cause uncontrolled tumor growth. The drug being used in this research study, ZD6474 (Vandetanib), is designed to block the receptors to two of these growth factors, the vascular endothelial growth factor (VEGF) and the epidermal growth factor (EGF). These growth factors are important in pathways that promote tumor growth and increasing blood supply to the tumor. Blocking these receptors may reduce the blood supply to the tumor and help slow down tumor growth. There is also laboratory evidence that blocking these receptors may increase the sensitivity of glioblastomas to radiation therapy.

This research study is a Phase I/II clinical trial.

Phase I clinical trials test the safety of an investigational drug. Phase I studies also try to define the appropriate dose of the investigational drug to use for further studies. We will determine the highest dose of ZD6474 (Vandetanib) that can be given safely when combined with temozolomide (Temodar) and radiation therapy.

The purpose of Phase II of this research study is to determine the efficacy of the combination treatment of ZD6474 (Vandetanib) with the standard therapy for glioblastomas and gliosarcomas, temozolomide (Temodar) and radiation therapy. It will look to see how patients fare on treatment (if they progress and when, how they are doing after 12 months of treatment). In this research study, the safety of the combination treatment of ZD6474 (Vandetanib) with the standard therapy for glioblastomas and gliosarcomas, temozolomide (Temodar) and radiation therapy will be further evaluated. We will also be looking at samples to see if there are correlations between them and how well patients do on treatment.

This agent is investigational for the treatment of glioblastomas. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it. It also means that the FDA (U.S. Food and Drug Administration) has not approved ZD6474 (Vandetanib) for use for your type of cancer. All subjects participating in this research study must NOT be taking a certain type of anti-seizure medication called enzyme inducing anticonvulsant drugs. These drugs include the following medications: Dilantin, Tegretol, Phenobarbital and trileptal.

ELIGIBILITY:
All inclusion and exclusion criteria apply to both phase I and II patients.

Inclusion Criteria:

* Subjects with histologically proven intracranial glioblastoma multiforme (GBM) and gliosarcoma will be eligible for this protocol.
* Gadolinium MRI or contrast CT must be obtained within 14 days prior to registration.
* Patients must have a plan to begin treatment with ZD6474 (vandetanib) and/or temozolomide 21 to 35 days after surgical resection or 14 to 35 days after stereotactic biopsy.
* Subjects must have a plan to begin partial brain radiotherapy 5-7 days after beginning ZD6474. Radiotherapy must be a) at the Radiation Oncology Department of the participating institution, b) at an affiliated site that is currently approved to participate in any trial of the Radiation Therapy Oncology Group (RTOG), or c) at another location with prior approval from the Overall PI of the trial. Radiotherapy must be given by external beam to a partial brain field in daily fractions of 180 to 200 cGy, to a planned total dose to the tumor of approximately 6000 cGy. Stereotactic radiosurgery and brachytherapy will not be allowed.
* If it is deemed in the best interest of the patient, intensity modulated radiation therapy (IMRT) is allowable on this trial. If IMRT is administered, dose specifics must be conducted per institutional guidelines.
* Subjects must be willing to forego other cytotoxic and non-cytotoxic drug therapy against the tumor while being treated with ZD6474 (ZactimaTM), with the exception of temozolomide.
* All subjects must sign an informed consent indicating that they are aware of the investigational nature of this study prior to any study-related procedures. Patients must be registered with in the Dana Farber Cancer Institute's Quality Assurance Office for Clinical Trials prior to treatment with ZD6474 (Vandetanib). Patients must sign an authorization for the release of their protected health information.
* Subjects can be male or female, and must be >/= 18 years old, with a life expectancy > 12 weeks.
* Subjects must be able to care for themselves (KPS>/=60).
* Subjects must have adequate labs as defined below:

  * Patients must have adequate bone marrow function (WBC >/= 3,000/μl, ANC >/= 1,500/mm3, platelet count of >/= 100,000/mm3, and hemoglobin >/= 10 gm/dl), adequate liver function (SGOT, SGPT </= 2.5 times ULN; bilirubin </= 1.5 times ULN), and adequate renal function (creatinine < 1.5 mg/dL, and/or serum creatinine </= 1.5 x ULN, and/or creatinine clearance > 30 mL/min, calculated by Cockcroft-Gault formula) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
  * Patients must have potassium >/= 4.0 mmol/L and serum calcium (ionized or adjusted for albumin) or magnesium in the normal range (supplementation is allowed).
  * Patients' alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be </= 2.5 X ULRR and their alkaline phosphatase (ALP) </= 2.5 x ULRR, (or </= 5x ULRR if judged by the investigator to be related to liver metastases)
* Women of childbearing potential must have a negative pregnancy test documented within 14 days prior to registration.
* Men and women of childbearing potential must agree to use adequate contraception while receiving study medication and continue for at least two months (five half-lives) after their last dose of study medication.
* Patients must have sufficient tissue available from their prior biopsy/surgery: at least 10 (preferably 20) unstained slides or 1 tissue block.
* Patients must agree not to donate blood during the trial and for 3 months following their last dose of trial treatment

Exclusion Criteria:

* Subjects must not have had prior cranial radiation therapy.
* Subjects must not have received prior cytotoxic drug therapy, non-cytotoxic drug therapy, or experimental drug therapy for brain tumors.
* Subjects must not have received prior Gliadel wafers.
* Subjects must not have received any investigational agents within 30 days prior to commencing study treatment
* Subjects must not have evidence of severe or uncontrolled systemic disease or any concurrent condition that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
* Subjects with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.
* Subjects must not have any unresolved toxicity greater than CTC grade 1 related to previous anti-cancer therapy.
* Subjects must not have active infection.
* Subjects must not be pregnant/breast feeding.
* Subjects must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Subjects must not have history of any clinically significant cardiac event, or evidence of heart disease.

  * No event such as myocardial infarction or superior vena cava syndrome (SVC); New York Heart Association (NYHA) classification of heart disease >/= 2 within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
  * No history of arrhythmia (multifocal premature ventricular contractions (PVCs), bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is not excluded.
  * No previous history of QTc prolongation as a result from other medication that required discontinuation of that medication.
  * No congenital long QT syndrome, or1st degree relative with unexplained sudden death under 40 years of age.
  * No left bundle branch block (LBBB).
  * Subject's screening ECG cannot indicate QTc (with Bazett's correction) that is either unmeasurable or >/= 480 msec on. If subject's screening QTc >/= 480 msec, it may be repeated twice (at least 24 hours apart). The average QTc from the 3 screening ECGs must be < 480 msec. Patients who are receiving a drug that has a risk of inducing Torsades de Pointes are excluded if QTc is >/= 460 msec.
* Subjects must not be taking any enzyme-inducing anti-epileptic drugs (EIAED) or other drugs that are potent inducers of CYP3A4 function (rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbitol and St. John's Wort). If patients were previously on EIAEDs and these have been discontinued, patients must have been off the agent for at least 7 days prior to registration.
* Subjects must not be taking concomitant medications known to prolong the QT interval and have a risk of inducing Torsade de Pointes (TdP). Any concurrent medication with a known risk of inducing TdP that, in the investigator's opinion cannot be discontinued, will be allowed; however, these patients must be monitored closely.
* Subjects must not have uncontrolled hypertension (high blood pressure).
* Subjects must not have active diarrhea that may affect the ability of the patient to absorb or tolerate ZD6474 (Vandetanib).
* Subjects with confirmed diagnosis of human immunodeficiency virus (HIV) infection are excluded at the investigator's discretion if he/she feels that 1) a potential drug interaction between ZD6474 (Vandetanib) and any of the patient's anti-HIV medications could influence the efficacy of the anti-HIV medication, or 2) it may place the patient at risk due to the pharmacologic activity of ZD6474 (Vandetanib).
* Subjects' pre-operative MRI must not demonstrate significant intratumoral or peritumoral hemorrhage & post-operative MRI must not demonstrate a large amount of peri-operative parenchymal hemorrhage. (Patients may have postoperative intracavitary blood.)
* Subjects must not have had major surgery (unrelated to the glioblastoma) within 4 weeks before starting study therapy, and subjects cannot have a surgical incision that has not completely healed before starting study therapy.
* Subjects must not be receiving Coumadin (subjects may take low molecular weight heparin).
* Subjects must not have enrolled on this trial previously.
* Subjects must have had no involvement in the planning or conduct of the study (applies to both AstraZeneca staff or staff at the study site).
* Any of the following lab results will result in patient exclusion from trial:

  * Potassium: < 4.0 mmol/L despite supplementation, or above the CTCAE grade 1 upper limit.
  * Magnesium below the normal range despite supplementation, or above the CTCAE grade 1 upper limit.
  * Serum calcium above the CTCAE grade 1 upper limit.

NOTE: In cases where the serum calcium is below the normal range, 2 options would be available:

* The calcium adjusted for albumin is to be obtained and substituted for the measured serum value. Exclusion is to then be based on the adjusted for albumin values falling below the normal limit.
* Determine the ionized calcium levels. If these ionized calcium levels are out of normal range despite supplementation, then the patient must be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-05-25 (Actual); Primary Completion 2013-08-31 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (7):
- United States (7):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber / Brigham and Women's Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 119 pts were registered & enrolled to trial, only 111 began study tx (8 enrolled pts did not receive tx on study). 7 pts randomized to Ph II Arm A removed their consent before starting study tx, and 1 Ph II Arm B pt was removed from study before starting tx, as pt clinically declined immediately following registration/randomization.
Groups:
- Phase I: Dose Level -1: RT + TMZ + Vandetanib @ 200 mg/Day; Phase I: Dose Level -2: RT + TMZ + Vandetanib @ 100 mg/Day: ZD6474 (Vandetanib) daily (to begin 5-7 days prior to starting participant's RT) Temozolomide (75 mg/m2 daily for 6 weeks) with concurrent fractionated radiation therapy for approximately 6 weeks (XRT must be given by external beam to a partial brain field in daily fractions of 180-200 cGy, to a planned total dose to the tumor of approximately 6000 cGy), followed by 4-6 weeks rest.
  Followed by:
  12 cycles of adjuvant temozolomide [at 150 mg/m2/day orally for 5 days (days 1-5) of a 28-day TMZ cycle; if 150 mg/m2/day is tolerated without difficulty and the investigator feels the patient can tolerate 200 mg/m2/day, then an increase to a maximum of 200 mg/m2/day for five days every 28 days may be given].
  ZD6474 (Vandetanib) daily for the twelve (12) 28-day cycles of adjuvant temozolomide, with the option to continue until participant experiences an unacceptable toxicity or his/her tumor progresses.
- Phase II: Arm B (Experimental Group: RT + TMZ + Vandetanib): The "Induction" Phase:
  ZD6474 (Vandetanib) daily (to begin 5-7 days prior to starting participant's RT) Temozolomide (75 mg/m2 daily for 6 weeks) with concurrent fractionated radiation therapy for approximately 6 weeks (XRT must be given by external beam to a partial brain field in daily fractions of 180-200 cGy, to a planned total dose to the tumor of approximately 6000 cGy), followed by 4-6 weeks rest.
  Followed by the "Maintenance" Phase:
  12 cycles of adjuvant temozolomide [at 150 mg/m2/day orally for 5 days (days 1-5) of a 28-day TMZ cycle; if 150 mg/m2/day is tolerated without difficulty and the investigator feels the patient can tolerate 200 mg/m2/day, then an increase to a maximum of 200 mg/m2/day for five days every 28 days may be given].
  ZD6474 (Vandetanib) daily for the twelve (12) 28-day cycles of adjuvant temozolomide, with the option to continue until participant experiences an unacceptable toxicity or his/her tumor progresses.
Period: Overall Study
Arm/Group | Phase I: Dose Level -1: RT + TMZ + Vandetanib @ 200 mg/Day | Phase I: Dose Level -2: RT + TMZ + Vandetanib @ 100 mg/Day | Phase II: Arm A (Control Group: RT + TMZ) | Phase II: Arm B (Experimental Group: RT + TMZ + Vandetanib)
Started | 6 | 7 | 29 | 69
Completed | 0 | 0 | 7 | 1
Not Completed | 6 | 7 | 22 | 68
Not completed — Adverse Event | 2 | 3 | 3 | 22
Not completed — Lack of Efficacy | 3 | 3 | 17 | 32
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 10
Not completed — Patient still receiving active study tx | 1 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level -1: RT + TMZ + Vandetanib @ 200 mg/Day | Phase I: Dose Level -2: RT + TMZ + Vandetanib @ 100 mg/Day | Phase II: Arm A (Control Group: RT + TMZ) | Phase II: Arm B (Experimental Group: RT + TMZ + Vandetanib) | Total
Number analyzed (Participants) | 6 | 7 | 29 | 69 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 24 | 50 | 85
  >=65 years | 0 | 2 | 5 | 19 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 13 | 25 | 41
  Male | 5 | 5 | 16 | 44 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 2 | 3
  White | 6 | 7 | 25 | 63 | 101
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 3 | 4
Baseline (Day 1) Karnofsky Performance Score (KPS) [Number; unit: Participants] — 100 Normal; no complaints/evidence of dz 90 Able to carry on normal activity; minor signs/symptoms of dz 80 Normal activity w/ effort; some sign/symptoms of dz 70 Cares for self; unable to carry on normal activity or do active work 60 Requires occasional assistance, but able to care for most personal needs 50 Requires considerable assistance & frequent medical care 40 Disabled; requires special care & assistance 30 Severely disabled; hosp indicated, although death not imminent 20 Very sick; hosp & active support tx necessary 10 Moribund; fatal processes progressing rapidly 0 Dead
  Participants
    100 | 0 | 5 | 7 | 15 | 27
    90 | 2 | 2 | 15 | 30 | 49
    80 | 1 | 0 | 2 | 17 | 20
    70 | 3 | 0 | 3 | 5 | 11
    60 | 0 | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced a Dose-limiting Toxicity (DLT)
Description: The primary outcome of Phase I of this trial was to determine the maximum tolerated dose (MTD) of ZD6474 (Vandetanib) in patients with newly-diagnosed glioblastomas multiforme (GBM) and gliosarcomas who are also receiving radiation therapy with concomitant and adjuvant temozolomide. The MTD is the dose level at which 0/6 or 1/6 patients experience a dose-limiting toxicity (DLT) with the next higher dose having at least 2/3 or 2/6 patients encountering DLT.
Time Frame: 2 years
Population: This measure was only assessed in Participants enrolled into the Phase I part of the study who had available data for analysis.
Measure: Number; unit: Participants
Arm/Group | Phase I: Dose Level -1: RT + TMZ + Vandetanib @ 200 mg/Day | Phase I: Dose Level -2: RT + TMZ + Vandetanib @ 100 mg/Day | Phase II: Arm A (Control Group: RT + TMZ) | Phase II: Arm B (Experimental Group: RT + TMZ + Vandetanib)
Number analyzed (Participants) | 6 | 6 | 0 | 0
Participants | 3 | 0 |  |

2. Primary Outcome: Median Overall Survival (OS) of Phase II Patients
Description: The primary outcome of Phase II of this trial was to determine the efficacy of ZD6474 (Vandetanib) in combination with radiation therapy and concomitant and adjuvant temozolomide in patients with newly-diagnosed GBM and gliosarcomas as measured by overall survival and median survival.
Time Frame: 3 years
Population: This measure was only assessed in Participants in Phase II part of the study, who had available data for analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: Dose Level -1: RT + TMZ + Vandetanib @ 200 mg/Day | Phase I: Dose Level -2: RT + TMZ + Vandetanib @ 100 mg/Day | Phase II: Arm A (Control Group: RT + TMZ) | Phase II: Arm B (Experimental Group: RT + TMZ + Vandetanib)
Number analyzed (Participants) | 0 | 0 | 29 | 69
months |  |  | 15.9 [11.0 to 22.5] | 16.6 [14.9 to 20.1]

3. Secondary Outcome: Median Progression-free Survival (PFS), as Calculated by the # of Months Patients Remain Progression-free
Description: A secondary outcome of Phase II of this trial is the median progression-free survival (PFS), as calculated by the # of months patients remain progression-free
Time Frame: 3 years
Population: This is an outcome for Phase II participants only; 0 Phase I participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I: Dose Level -1: RT + TMZ + Vandetanib @ 200 mg/Day | Phase I: Dose Level -2: RT + TMZ + Vandetanib @ 100 mg/Day | Phase II: Arm A (Control Group: RT + TMZ) | Phase II: Arm B (Experimental Group: RT + TMZ + Vandetanib)
Number analyzed (Participants) | 0 | 0 | 29 | 69
months |  |  | 6.2 [3.9 to 10.4] | 7.7 [5.5 to 10.1]

4. Secondary Outcome: PHASE II: Percentage of Grade 3-5 Treatment-Related Adverse Events
Description: The percentage of adverse events (based on CTCAEv3) reported on study (via case report forms and Reportable AE submissions) that are both high-grade (grade 3, 4, or 5) and considered at least possibly related to study treatment.
Time Frame: Adverse events experienced by participants are collected and reported throughout treatment with study drug (from initiation of study treatment until 30 days after the last dose of study treatment), maximum timeframe was 6 years.
Measure: Number (95% Confidence Interval); unit: percentage of events
Groups:
- Phase II - Arm A - Participants: Phase II Control Arm: Arm A (RT + TMZ)
- Phase II - Arm B - Participants: Phase II Treatment Arm: Arm B (RT + TMZ + Vandetanib)
Arm/Group | Phase II - Arm A - Participants | Phase II - Arm B - Participants
Number analyzed (Participants) | 29 | 69
percentage of events | 4.16 [2.56 to 6.35] | 8.37 [6.85 to 10.10]

5. Secondary Outcome: PHASE I: Percentage of Grade 3-5 Treatment-Related Adverse Events
Description: as for outcome 4
Time Frame: Adverse events experienced by participants are collected and reported throughout treatment with study drug (from initiation of study treatment until 30 days after the last dose of study treatment), maximum timeframe was 7 years.
Measure: Number (95% Confidence Interval); unit: percentage of events
Groups:
- Phase I Participants - Vandetanib @ 200 mg/Day: Phase I Participants (RT + TMZ + Vandetanib): Cohorts 1 & 2 (Vandetanib @ 200 mg/day)
- Phase I Participants - Vandetanib @ 100 mg/Day: Phase I Participants (RT + TMZ + Vandetanib): Cohorts 3 & 4 (Vandetanib @ 100 mg/day)
Arm/Group | Phase I Participants - Vandetanib @ 200 mg/Day | Phase I Participants - Vandetanib @ 100 mg/Day
Number analyzed (Participants) | 6 | 7
percentage of events | 9.48 [5.15 to 15.68] | 4.43 [1.8 to 8.92]

ADVERSE EVENTS:
Time Frame: AEs & SAEs are collected from consent throughout tx period, including a follow-up period (30 days after last dose or until resolution). All study-related AEs are followed until resolution, unless deemed by the Investigator unlikely to resolve.
Description: Although 29 pts received study tx in the Phase II - Arm A group, the # of pts at risk for SAEs in the "Phase II-Arm A Pts (Control Group): RT + TMZ" group is reported as 30 to include 1 additional Arm A pt who did not ultimately start study tx who experienced a Reportable AE (gr3 confusion w/ urinary incontinence) on the date pt was registered.
Groups:
- Phase I & Phase II-Arm B Pts: RT + TMZ + Vandetanib: The "Induction" Phase:
  ZD6474 (Vandetanib) daily (to begin 5-7 days prior to starting participant's RT) Temozolomide (75 mg/m2 daily for 6 weeks) with concurrent fractionated radiation therapy for approximately 6 weeks (XRT must be given by external beam to a partial brain field in daily fractions of 180-200 cGy, to a planned total dose to the tumor of approximately 6000 cGy), followed by 4-6 weeks rest.
  Followed by the "Maintenance" Phase:
  12 cycles of adjuvant temozolomide [at 150 mg/m2/day orally for 5 days (days 1-5) of a 28-day TMZ cycle; if 150 mg/m2/day is tolerated without difficulty and the investigator feels the patient can tolerate 200 mg/m2/day, then an increase to a maximum of 200 mg/m2/day for five days every 28 days may be given].
  ZD6474 (Vandetanib) daily for the twelve (12) 28-day cycles of adjuvant temozolomide, with the option to continue until participant experiences an unacceptable toxicity or his/her tumor progresses.
- Phase II-Arm A Pts (Control Group): RT + TMZ: The "Induction" Phase:
  Temozolomide (75 mg/m2 daily for 6 weeks) with concurrent fractionated radiation therapy for approximately 6 weeks (XRT must be given by external beam to a partial brain field in daily fractions of 180-200 cGy, to a planned total dose to the tumor of approximately 6000 cGy), followed by 4-6 weeks rest.
  Followed by the "Maintenance" Phase:
  12 cycles of adjuvant temozolomide [at 150 mg/m2/day orally for 5 days (days 1-5) of a 28-day TMZ cycle; if 150 mg/m2/day is tolerated without difficulty and the investigator feels the patient can tolerate 200 mg/m2/day, then an increase to a maximum of 200 mg/m2/day for five days every 28 days may be given].
Arm/Group | Phase I & Phase II-Arm B Pts: RT + TMZ + Vandetanib | Phase II-Arm A Pts (Control Group): RT + TMZ
Serious Adverse Events (participants affected / at risk) | 52/82 | 15/30
Other Adverse Events (participants affected / at risk) | 81/82 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I & Phase II-Arm B Pts: RT + TMZ + Vandetanib (N=82) | Phase II-Arm A Pts (Control Group): RT + TMZ (N=30)
hemoglobin (Blood and lymphatic system disorders) | 2 | 1
lymphopenia (Blood and lymphatic system disorders) | 8 | 1
neutrophils (Blood and lymphatic system disorders) | 7 | 3
platelets (Blood and lymphatic system disorders) | 4 | 4
leukocytes (Blood and lymphatic system disorders) | 0 | 0
blood/bone marrow: other: hemolytic anemia (Blood and lymphatic system disorders) | 1 | 0
fatigue (General disorders) | 1 | 1
fever without neutropenia (General disorders) | 3 | 1
supraventricular and nodal arrhythmia: atrial fibrillation (Cardiac disorders) | 1 | 0
hypertension (Cardiac disorders) | 1 | 0
hypotension (Cardiac disorders) | 1 | 0
death - disease progression (General disorders) | 1 | 0
death NOS (General disorders) | 1 | 0
erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
wound - non-infectious (Skin and subcutaneous tissue disorders) | 1 | 0
adrenal insufficiency (Endocrine disorders) | 0 | 1
anorexia (Gastrointestinal disorders) | 0 | 1
ascites (non-malignant) (Gastrointestinal disorders) | 1 | 0
dehydration (Gastrointestinal disorders) | 0 | 1
diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 0
duodenum, hemorrhage (Gastrointestinal disorders) | 1 | 0
fistula, colon/cecum/appendix (Gastrointestinal disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0
perforation, colon (Gastrointestinal disorders) | 2 | 0
stomach, hemorrhage (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 0
CNS, hemorrhage (Nervous system disorders) | 1 | 0
hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hematoma (Vascular disorders) | 0 | 1
cholecystitis (Hepatobiliary disorders) | 1 | 0
liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 | 0
infection gr0-2 neut, appendix (Infections and infestations) | 1 | 0
infection gr0-2 neut, lung (Infections and infestations) | 3 | 0
infection gr0-2 neut, nose (Infections and infestations) | 1 | 0
infection gr0-2 neut, skin (Infections and infestations) | 1 | 0
infection gr0-2 neut, urinary tract (Infections and infestations) | 1 | 2
infection gr0-2 neut, wound (Infections and infestations) | 1 | 0
infection w/ gr3-4 neut, wound (Infections and infestations) | 1 | 0
infection gr0-2 neut, anal/perianl (Infections and infestations) | 0 | 1
infection: other: eye infection (Infections and infestations) | 0 | 1
infection: other: infection of the leg (Infections and infestations) | 1 | 0
edema: head and neck (cerebral edema) (General disorders) | 1 | 0
ALT, SGPT (Metabolism and nutrition disorders) | 3 | 0
AST, SGOT (Metabolism and nutrition disorders) | 3 | 0
bilirubin (Metabolism and nutrition disorders) | 1 | 0
hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
metabolic/laboratory: other: immunosupression (Metabolism and nutrition disorders) | 1 | 0
nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
nonneuropathic left-side muscle weak (Musculoskeletal and connective tissue disorders) | 1 | 0
musculoskeletal/soft tissue: other: steroid myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 0 | 1
musculoskeletal/soft tissue: other: bulging discs (Musculoskeletal and connective tissue disorders) | 0 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0
confusion (Nervous system disorders) | 1 | 2
dizziness (Nervous system disorders) | 1 | 0
mental status (Nervous system disorders) | 1 | 0
neuropathy-motor (Nervous system disorders) | 1 | 0
neuropathy-sensory (Nervous system disorders) | 1 | 0
neurology: other: vasogenic cerebral edema (Nervous system disorders) | 1 | 0
seizure (Nervous system disorders) | 6 | 2
speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 2 | 1
syncope (fainting) (Nervous system disorders) | 1 | 0
cognitive disturbance (Nervous system disorders) | 0 | 1
vision-blurred (Eye disorders) | 1 | 0
pain - chest/thorax NOS (General disorders) | 1 | 0
pain - head/headache (Nervous system disorders) | 1 | 0
pain - abdomen NOS (Gastrointestinal disorders) | 2 | 0
pain - muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
pain - throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
obstruction, airway-bronchus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
obstruction-ureteral (Renal and urinary disorders) | 1 | 0
renal failure (Renal and urinary disorders) | 1 | 0
urinary retention (Renal and urinary disorders) | 2 | 1
incontinence, urinary (Renal and urinary disorders) | 0 | 1
thrombosis/thrombus/embolism (Vascular disorders) | 18 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I & Phase II-Arm B Pts: RT + TMZ + Vandetanib (N=82) | Phase II-Arm A Pts (Control Group): RT + TMZ (N=29)
hemoglobin (Blood and lymphatic system disorders) | 38 | 19
leukocytes (Blood and lymphatic system disorders) | 34 | 12
lymphopenia (Blood and lymphatic system disorders) | 43 | 16
neutrophils (Blood and lymphatic system disorders) | 21 | 9
platelets (Blood and lymphatic system disorders) | 48 | 13
blood/bone marrow: other: decreased hematocrit (Blood and lymphatic system disorders) | 6 | 1
blood/bone marrow: other: decreased red blood cells (Blood and lymphatic system disorders) | 3 | 2
blood/bone marrow: other: increase eosinophils (Blood and lymphatic system disorders) | 2 | 2
PTT (Investigations) | 5 | 1
fatigue (General disorders) | 62 | 22
insomnia (Psychiatric disorders) | 20 | 1
weight loss (Investigations) | 7 | 2
alopecia (Skin and subcutaneous tissue disorders) | 18 | 6
chemoradiation dermatitis (Skin and subcutaneous tissue disorders) | 5 | 2
erythema multiforme (Skin and subcutaneous tissue disorders) | 6 | 0
pruritus/itching (Skin and subcutaneous tissue disorders) | 7 | 0
rash/desquamation (Skin and subcutaneous tissue disorders) | 23 | 2
rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 17 | 3
dry skin (Skin and subcutaneous tissue disorders) | 4 | 3
radiation dermatitis (Skin and subcutaneous tissue disorders) | 3 | 4
cushingnoid appearance (Endocrine disorders) | 5 | 5
adrenal insufficiency (Endocrine disorders) | 0 | 2
anorexia (Gastrointestinal disorders) | 16 | 9
constipation (Gastrointestinal disorders) | 17 | 9
diarrhea w/o prior colostomy (Gastrointestinal disorders) | 25 | 2
dyspepsia (Gastrointestinal disorders) | 9 | 2
nausea (Gastrointestinal disorders) | 33 | 11
taste disturbance (Gastrointestinal disorders) | 6 | 1
vomiting (Gastrointestinal disorders) | 17 | 4
dehydration (Gastrointestinal disorders) | 2 | 2
infection gr0-2 neut, oral cavity (Infections and infestations) | 5 | 3
infection gr0-2 neut, conjunctiva (Infections and infestations) | 0 | 3
infection gr0-2 neut, upper airway (Infections and infestations) | 3 | 2
infection gr0-2 neut, urinary tract (Infections and infestations) | 4 | 3
hemorrhage, pulmonary/upper respiratory: nose (Respiratory, thoracic and mediastinal disorders) | 3 | 2
edema, head and neck (General disorders) | 0 | 3
edema, limb (General disorders) | 10 | 5
alkaline phosphatase (Metabolism and nutrition disorders) | 11 | 3
ALT, SGPT (Metabolism and nutrition disorders) | 48 | 15
AST, SGOT (Metabolism and nutrition disorders) | 37 | 10
bicarbonate (Metabolism and nutrition disorders) | 17 | 8
bilirubin (Metabolism and nutrition disorders) | 17 | 4
creatinine (Metabolism and nutrition disorders) | 18 | 2
hypercalcemia (Metabolism and nutrition disorders) | 7 | 1
hyperglycemia (Metabolism and nutrition disorders) | 50 | 19
hyperkalemia (Metabolism and nutrition disorders) | 18 | 5
hypermagnesemia (Metabolism and nutrition disorders) | 7 | 4
hypernatremia (Metabolism and nutrition disorders) | 6 | 2
hypoalbuminemia (Metabolism and nutrition disorders) | 19 | 3
hypocalcemia (Metabolism and nutrition disorders) | 19 | 4
hypoglycemia (Metabolism and nutrition disorders) | 17 | 2
hypokalemia (Metabolism and nutrition disorders) | 17 | 7
hypomagnesemia (Metabolism and nutrition disorders) | 6 | 4
hyponatremia (Metabolism and nutrition disorders) | 25 | 5
hypophosphatemia (Metabolism and nutrition disorders) | 22 | 7
proteinuria (Metabolism and nutrition disorders) | 17 | 5
hyperuricemia (Metabolism and nutrition disorders) | 0 | 2
metabolic/laboratory: other: elevated BUN (Metabolism and nutrition disorders) | 3 | 2
metabolic/laboratory: other: hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 2
extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 5 | 2
nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 9 | 2
nonneuropathic left-side muscle weak (Musculoskeletal and connective tissue disorders) | 5 | 1
nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 8 | 2
anxiety (Nervous system disorders) | 14 | 4
ataxia (Nervous system disorders) | 7 | 3
cognitive disturbance (Nervous system disorders) | 6 | 6
confusion (Nervous system disorders) | 14 | 4
depression (Nervous system disorders) | 19 | 2
dizziness (Nervous system disorders) | 15 | 6
memory impairment (Nervous system disorders) | 20 | 7
neuropathy CN II vision (Nervous system disorders) | 6 | 0
neuropathy-motor (Nervous system disorders) | 7 | 2
neuropathy-sensory (Nervous system disorders) | 11 | 4
seizure (Nervous system disorders) | 11 | 5
speech impairment (Nervous system disorders) | 8 | 6
tremor (Nervous system disorders) | 12 | 4
personality (Nervous system disorders) | 0 | 2
vision - blurred (Eye disorders) | 6 | 3
pain, abdomen, NOS (Gastrointestinal disorders) | 6 | 2
pain, back (Musculoskeletal and connective tissue disorders) | 5 | 4
pain, extremity-limb (Musculoskeletal and connective tissue disorders) | 6 | 1
pain, head/headache (Nervous system disorders) | 29 | 16
pain, joint (Musculoskeletal and connective tissue disorders) | 5 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 17 | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
urinary frequency/urgency (Renal and urinary disorders) | 11 | 4
incontinence urinary (Renal and urinary disorders) | 4 | 3
thrombosis/thrombus/embolism (Vascular disorders) | 18 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days